CLINICAL TRIAL: NCT03331991
Title: Prevention of Influenza and Other Wintertime Respiratory Viruses Among Healthcare Professionals in Israel
Acronym: HCP
Status: Completed | Type: Observational
Sponsor: Abt Associates (Industry)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Clalit Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HHSD2002013M53890B
Record Dates: First submitted 2016-07-27; First posted 2017-11-06 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2017-11

CONDITIONS: Respiratory Tract Disease; Influenza
MeSH Terms: conditions — Respiratory Tract Diseases; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens and respiratory specimens will be collected.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: influenza vaccine — exposure to influenza vaccine

SUMMARY:
The purpose of the study on the Prevention of Influenza and Other Wintertime Respiratory Viruses among Healthcare Professionals in Israel Effectiveness of Influenza Vaccine in Preventing Influenza Virus Infection, Missed Work, and Patient Exposure: A Prospective Cohort Study of Healthcare Personnel (to be called the Healthcare Personnel or HCP study throughout this Data Security Plan) is to investigate vaccine effectiveness and respiratory illness among healthcare personnel (HCP). This will help to better understand the factors that influence influenza vaccination choice, individual vaccine response, and whether or not the influenza vaccine helps to prevent influenza in HCP.

DETAILED DESCRIPTION:
Healthcare personnel (HCP) are believed to be at increased risk of influenza infection and often work while ill, which increases the risk of secondary exposure to vulnerable patients. Vaccination of HCP against influenza is an important component of infection control in healthcare settings, but persistently low rates of vaccine uptake among HCP remains a topic of international concern and debate. Although recent reviews confirm that the seasonal influenza vaccine is moderately effective in reducing the risk of influenza illness [10], multiple gaps in knowledge remain regarding the preventive value of vaccine among HCP.

During at least two consecutive influenza seasons or years, this prospective cohort study of healthcare personnel in middle-income countries has four primary objectives: (1) Describe the frequency and impact of acute respiratory illnesses (ARI) among HCP during wintertime; (2) Estimate the effectiveness of influenza vaccine in preventing symptomatic influenza illness, missed work due to influenza illness, and hours of direct patient care provided by HCP with symptomatic influenza infections; (3) Examine the association between repeated influenza vaccination and HCP's baseline immune landscape, their response to influenza vaccines, and their subsequent protection against infection; (4) Examine if influenza vaccine modifies symptom severity and duration among HCP with breakthrough influenza infections despite vaccination.

Approximately 2,400-2,800 HCP providing direct patient care will be enrolled in a prospective cohort to be followed for at least two years (or two influenza seasons). In Israel, approximately 1,200 HCPs will be enrolled in Year 1 of the study, with an expansion to full enrollment in Year 2. Thus, the investigators anticipate a 3 year cohort study in which ~1,200 participants will contribute to years 1 and 2 of the study and the remaining sample will contribute to years 2 and 3 of the study. Information on socio-demographic characteristics, current medical conditions, medical history, medical care utilization, and influenza vaccination history will be extracted from medical and employee records with the participant's permission. Other information on socio-demographics, occupational responsibilities, health status, and knowledge and attitudes about viruses and vaccines will be collected by self-report through an enrollment survey. Collection of blood specimens will occur prior to and after influenza seasons during each study year; in addition, HCP who receive the influenza vaccine will provide an additional blood draw 21-42 days after vaccination. Active surveillance to identify acute illnesses (associated with cough, runny nose, body aches, or feverishness) will occur twice-weekly during weeks of local influenza circulation. When an acute illness is identified, participants will provide a respiratory specimen (nasal self-swab) for influenza testing and complete two brief surveys during and after resolution of their illness. For a sub-sample of consented participants, additional information on attitudes toward morbidity with influenza and respiratory illness will be collected through in-depth qualitative interviews. Additional brief surveys will be completed at the end of each season/year and at the start of the second influenza season to update information on participant health, work responsibilities, and attitudes and practices associated with vaccination and other inflection control and prevention measures.

ELIGIBILITY:
Inclusion Criteria:

* Be aged ≥18 years old;
* Work at the facility full-time (≥30 hours per week);
* Have routine direct hands-on or face-to-face contact with patients (within 1 meter) as part of a typical work shift, including, but not limited to, physicians, nurses, respiratory therapists, physical therapists, unit clerks, radiograph technicians, medical assistants, and transporters;
* Continuous membership in Clalit Health plan for at least 1 year prior to enrollment.

Exclusion Criteria:

* No routine direct patient contact;
* Works part-time;
* Already received current season's flu vaccine more than 48 hours before enrollment and, thus, cannot complete blood draw prior to full immune response to the vaccine;
* Not be a member of the Clalit Health System health plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare personnel
Sampling Method: Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Frequency of acute respiratory illness among healthcare personnel receiving influenza vaccine | 3 years
Proportion of work days missed associated with self-reported acute respiratory illness | 3 years

SECONDARY OUTCOMES:
Frequency of asymptomatic and symptomatic infections (with typical or atypical symptom manifestations) with influenza viruses (and other viruses) | 3 years
Knowledge, attitudes, and practices (KAP) that predict vaccination hesitancy and refusal among healthcare personnel | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Thompson, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Rabin Medical Center, Petah Tikva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirsch A, Katz MA, Laufer Peretz A, Greenberg D, Wendlandt R, Shemer Avni Y, Newes-Adeyi G, Gofer I, Leventer-Roberts M, Davidovitch N, Rosenthal A, Gur-Arie R, Hertz T, Glatman-Freedman A, Monto AS, Azziz-Baumgartner E, Ferdinands JM, Martin ET, Malosh RE, Neyra Quijandria JM, Levine M, Campbell W, Balicer R, Thompson MG; SHIRI workgroup. Study of Healthcare Personnel with Influenza and other Respiratory Viruses in Israel (SHIRI): study protocol. BMC Infect Dis. 2018 Nov 6;18(1):550. doi: 10.1186/s12879-018-3444-7. PMID 30400834